CLINICAL TRIAL: NCT04076943
Title: A Phase 2 Open Label Study Investigating the Efficacy and Safety of Roxadustat (FG-4592) for Treatment of Anemia in Patients Receiving Chemotherapy Treatment for Non-Myeloid Malignancies
Brief Title: Evaluation of Efficacy and Safety of Roxadustat for the Treatment of Chemotherapy Induced Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: AstraZeneca (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-092
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Results first posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Chemotherapy Induced Anemia
Keywords: Anemia; Chemotherapy induced anemia; Myelosuppressive chemotherapy; Non-Myeloid malignances
MeSH Terms: conditions — Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Roxadustat (Experimental): Participants will receive roxadustat as an oral tablet, 3 times per week (TIW) for up to a maximum of 16 weeks.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Roxadustat will be administered per schedule specified in the arm description.
  Other Names: FG-4592

SUMMARY:
The purpose of this study is to find out if roxadustat (also known as FG-4592) is safe and effective for the treatment of anemia in participants receiving chemotherapy treatment for cancer.

DETAILED DESCRIPTION:
This study consists of three periods:

1. Screening Period up to 28 days
2. Treatment Period of up to16 weeks
3. A Follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of non-myeloid malignancy
2. Anemia caused by cancer treatment (myelosuppressive chemotherapy) defined as Hb ≤10.0 grams (g)/deciliter (dL) at screening
3. Planned concurrent treatment of cancer with chemotherapy for at least 8 additional weeks
4. Estimated life expectancy ≥ 6 months at enrollment (Day 1)

Exclusion Criteria:

1. Participants with cancer receiving chemotherapy when the anticipated outcome is cure
2. Participants who are only receiving hormonal products, biological products, cancer immunotherapy or radiation therapy to treat/manage their cancer
3. History of leukemia
4. Participants who have received an RBC transfusion or erythropoietic therapy within 4 weeks of enrollment
5. Use of any investigational drug within 8-weeks prior to treatment with roxadustat
6. Clinically significant anemia due to other etiologies
7. Cardiovascular risks, such as myocardial infarction, stroke, heart failure or thromboembolic event (for example, deep vein thrombosis [DVT] or pulmonary embolism) within previous 6 months of screening
8. Clinically significant or uncontrolled ongoing autoimmune disease (for example, rheumatoid arthritis, Crohn's disease, celiac disease, etc.)
9. Known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Research Center, Los Alamitos, California
  - Research Center, Los Angeles, California
  - Research Center, Torrance, California
  - Research Center, Jacksonville, Florida
  - Research Center, Plantation, Florida
  - Research Center, Fort Wayne, Indiana
  - Research Center, Ashland, Kentucky
  - Research Center, Covington, Louisiana
  - Research Center, Bethesda, Maryland
  - Research Center, Livingston, New Jersey
  - Research Center, Port Jefferson Station, New York
  - Research Center, The Bronx, New York
  - Research Center, Canton, Ohio
  - Research Center, Gettysburg, Pennsylvania
  - Research Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Roxadustat: Participants received roxadustat as an oral tablet, 3 times per week (TIW) for up to a maximum of 16 weeks. The starting dose of roxadustat was 2.0 milligrams (mg)/kilogram (kg). The dose was updated with Amendment 3 (dated 22 May 2020) for newly enrolled participants by 1 level that is, from 2.0 mg/kg to 2.5 mg/kg level to achieve an improved hemoglobin (Hb) response.
Period: Overall Study
Arm/Group | Roxadustat
Started | 92
Received at Least 1 Dose of Study Drug | 92
Completed | 58
Not Completed | 34
Not completed — Withdrawal by Subject | 12
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 2
Not completed — Death | 13
Not completed — Other than specified | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants enrolled in the roxadustat treatment period and received at least 1 dose of study medication.
Groups:
- Roxadustat: Participants received roxadustat as an oral tablet, TIW for up to a maximum of 16 weeks. The starting dose of roxadustat was 2.0 mg/kg. The dose was updated with Amendment 3 (dated 22 May 2020) for newly enrolled participants by 1 level that is, from 2.0 mg/kg to 2.5 mg/kg level to achieve an improved Hb response.
Arm/Group | Roxadustat
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 76
  Black or African American | 12
  Asian | 3
  Other | 1
Baseline Hemoglobin (Hb) [Mean (Standard Deviation); unit: grams (g)/deciliter (dL)] | 8.59 (0.956)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change in Hb Within 16 Weeks From Baseline Without Red Blood Cell (RBC) Transfusion
Description: Baseline Hb was defined as the mean of the assessments from central lab prior to first dose of the study treatment, which included up to 2 latest screening values prior to Day 1 and a value on Day 1. All central lab assessments from Day 1 to end of treatment (EOT) or early termination (ET) were included in the evaluation of this endpoint. Hb values within 4 weeks after an RBC transfusion were excluded.
Time Frame: Baseline, up to Week 16
Population: Full analysis set included all enrolled participants who received at least 1 dose of roxadustat, had a baseline Hb and at least 1 central lab Hb assessment during the treatment period.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat
Number analyzed (Participants) | 89
g/dL | 2.47 (1.510)

2. Secondary Outcome: Mean Change in Hb Level From Baseline to Week 16 (Without RBC Transfusion)
Description: Baseline Hb was defined as the mean of the assessments from central lab prior to first dose of the study treatment, which included up to 2 latest screening values prior to Day 1 and a value on Day 1. Mean Hb during treatment was computed using the mean area-under-the-curve trapezoid method, from Day 1 to EOT or ET Hb assessment.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat
Number analyzed (Participants) | 89
g/dL | 1.20 (1.012)

3. Secondary Outcome: Change in Hb From Baseline at Weeks 9, 13, and 16 (Without RBC Transfusion)
Description: Baseline Hb was defined as the mean of the assessments from central lab prior to first dose of the study treatment, which included up to 2 latest screening values prior to Day 1 and a value on Day 1.
Time Frame: Baseline, Weeks 9, 13, and 16
Population: Full analysis set included all enrolled participants who received at least 1 dose of roxadustat, had a baseline Hb and at least 1 central lab Hb assessment during the treatment period. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat
Number analyzed (Participants) | 61
g/dL
  Change at Week 9 | 1.43 (1.421)
  Change at Week 13: number analyzed (Participants) | 51
  Change at Week 13 | 2.15 (1.921)
  Change at Week 16: number analyzed (Participants) | 51
  Change at Week 16 | 2.52 (1.700)

4. Secondary Outcome: Percentage of Participants Who Achieved a ≥1 g/dL Increase in Hb From Baseline Through Week 16
Description: The 95% confidence interval (CI) was based on the exact method of Clopper-Pearson method. All central lab assessments from Day 1 to EOT or ET were included in the analysis. Hb values within 4 weeks after an RBC transfusion was excluded.
Time Frame: Baseline through Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 89
percentage of participants | 82.0 [72.5 to 89.4]

5. Secondary Outcome: Time to Achieve a ≥1 g/dL Increase in Hb From Baseline Through Week 16
Description: Median was calculated using Kaplan-Meier product limit method. 95% CI was calculated using the method of Brookmeyer and Crowley. All central lab assessments from Day 1 to EOT or ET were included in the analysis. Hb values within 4 weeks after an RBC transfusion were excluded.
Time Frame: Baseline through Week 16
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Roxadustat
Number analyzed (Participants) | 89
days | 41.0 [29.0 to 46.0]

6. Secondary Outcome: Percentage of Participants Who Achieved a ≥1.5 g/dL Increase in Hb From Baseline Through Week 16
Description: The 95% CI was based on the exact method of Clopper-Pearson method. All central lab assessments from Day 1 to EOT or ET were included in the analysis. Hb values within 4 weeks after an RBC transfusion was excluded.
Time Frame: Baseline through Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 89
percentage of participants | 73.0 [62.6 to 81.9]

7. Secondary Outcome: Percentage of Participants Who Achieved a Hematopoietic Response
Description: Hematopoietic response was defined as an increase in Hb of 1.5 g/dL from baseline or attaining a Hb of 11 g/dL. The 95% CI was based on the exact method of Clopper-Pearson method. All central lab assessments from Day 1 to EOT or ET were included in the analysis. Hb values within 4 weeks after an RBC transfusion was excluded.
Time Frame: Baseline through Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 89
percentage of participants | 75.3 [65.0 to 83.8]

8. Secondary Outcome: Percentage of Participants Who Achieved a ≥2 g/dL Increase in Hb From Baseline Through Week 16
Description: as for outcome 6
Time Frame: Baseline through Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 89
percentage of participants | 60.7 [49.7 to 70.9]

9. Secondary Outcome: Percentage of Participants Who Had an RBC Transfusion From Beginning of Week 5 (Day 29) to Week 16
Time Frame: Week 5 to Week 16
Population: Full analysis set included all enrolled participants who received at least 1 dose of roxadustat, had a baseline Hb and at least 1 central lab Hb assessment during the treatment period. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Roxadustat
Number analyzed (Participants) | 83
percentage of participants | 14.5

ADVERSE EVENTS:
Time Frame: Baseline up to Week 20
Description: Safety population included all participants who took at least 1 dose of study medication.
Arm/Group | Roxadustat
All-Cause Mortality (participants affected / at risk) | 17/92
Serious Adverse Events (participants affected / at risk) | 40/92
Other Adverse Events (participants affected / at risk) | 71/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=92)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Chills (General disorders) | 1
Disease progression (General disorders) | 3
COVID-19 pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Retroperitoneal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 2
Status epilepticus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Bladder pain (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Anoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Vena cava embolism (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=92)
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 23
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 6
Fall (Injury, poisoning and procedural complications) | 5
Decreased appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 6
Deep vein thrombosis (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT04076943/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04076943/SAP_001.pdf